CLINICAL TRIAL: NCT00183222
Title: Alcohol Research Center Grant. Component #1. COMBINING MEDICATIONS: ALCOHOL REACTIVITY AND CONSUMPTION
Brief Title: Effectiveness of Naltrexone and/or Ondansetron to Reduce Craving for Alcohol and Drinking
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: NIAAAANT010761-2005a; P50AA010761 (NIH); NIH Grant P50 AA010761
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2010-05-05 (Estimated); Status verified 2010-05

CONDITIONS: Alcohol Dependence
Keywords: Alcohol dependence; Alcoholism; Craving
MeSH Terms: conditions — Alcoholism | interventions — Naltrexone; Ondansetron; WW Domain-Containing Oxidoreductase

INTERVENTIONS:
Drug: naltrexone (up to 50 mg/day) for 8 days; ondansetron (0.25 mg twice a day) for 8 days

SUMMARY:
The purpose of this study is to determine whether naltrexone (an opiate blocking agent approved for the treatment of alcohol dependence), ondansetron a serotonin 3 antagonist medication approved to treat nausea) or their combination are effective in the reduction of alcohol craving and drinking compared to placebo.

DETAILED DESCRIPTION:
Non-treatment seeking individuals meeting criteria for alcohol dependence N=160) will be recruited through advertisement and paid for their participation. Alcoholics, after baseline evaluation, will be assigned through urn randomization (using a double dummy placebo controlled design) to one of four experimental groups, naltrexone (50 mg/day) (N=40), ondansetron (0.25 mg twice a day) (N=40), naltrexone and ondansetron (N=40) or placebos (N=40). Subjects will take the study drugs for 8 days (day 1-5 being the natural observation period). After a minimum of 48 hours of abstinence from alcohol day 6-8) they will undergo an alcohol administration (priming dose) and motivated free choice drinking procedure (on day 8). Alcoholic subjects will receive a brief counseling session at the end of the study to enhance their awareness of problem drinking and to motivate them to seek treatment. Referral for treatment will be offered.A subset of subjects from each medication group (N=15) will undergo a functional MRI brain scan with cue stimulation on day 7, on the evening before the alcohol administration paradigm.

A smaller group of social drinker controls (N=16), recruited and paid in a similar fashion, will be randomly assigned to the same medication groups (4 per group). They will be used as procedure controls for the alcohol administration lab study and as a comparison/contrast group for the brain imaging sub-study.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria (alcohol dependent group):

1. Age 21 65
2. Meets the DSM IV criterion for current alcohol dependence including "loss of control over drinking" (criterion 4) but does not necessarily have signs of physiologic dependence as expressed in criterion for tolerance development (criterion 1) and withdrawal symptoms or use to avoid withdrawal symptoms (criterion 2).
3. Currently is not engaged in, and does not want treatment for, alcohol related problems.
4. Able to read and understand questionnaires and informed consent.
5. Lives within 50 miles of the study site.
6. Able to maintain abstinence for up to three days (without the aid of detox medications) as determined by self report and breathalyzer measurements.

Inclusion Criteria (social drinker group):

1. Age 21 65
2. Does not meet the DSM IV criterion for lifetime or current alcohol abuse or dependence.
3. Consumes, on average, less than 14 standard drinks per week. But has consumed at least 2 standard drinks on at least one occasion in the last month.
4. Currently is not engaged in, and does not want, treatment for alcohol related problems.
5. Able to read and understand questionnaires and informed consent.
6. Able to maintain abstinence for three days.

Inclusion for fMRI imaging sub-study (see methodology section for rationale):

1. Does not have metal objects in the head/neck.
2. Does not have a history of claustrophobia leading to significant clinical anxiety symptoms.
3. Between the age of 25-45 years.
4. Does not currently smoke (note: 62% of our current sample are non-smokers).

Exclusion Criteria:

1. Currently meets DSM IV criteria for any other psychoactive substance dependence disorder.
2. History of opiate abuse or a positive urine drug screen for opiates.
3. Any psychoactive substance use (except marijuana and nicotine) within the last 30 days as evidenced by self-report and urine drug screen. For marijuana -no use within the last seven days.
4. Meets DSM IV criteria for current axis I disorders of major depression, panic disorder, obsessive compulsive disorder, post traumatic stress syndrome, bipolar affective disorder, schizophrenia, dissociate disorders and eating disorders, any other psychotic disorder or organic mental disorder.
5. Has current suicidal ideation or homicidal ideation.
6. Need for maintenance or acute treatment with any psychoactive medication including anti-seizure medications.
7. Current use of disulfiram.
8. Clinically significant medical problems such as, cardiovascular, renal, GI, or endocrine problem that would impair participation or limit medication ingestion.
9. Past history of alcohol related medical illness such as gastrointestinal bleeding, pancreatitis, peptic ulcer, hepatic cirrhosis or alcoholic hepatitis.
10. Hepatocellular disease indicated by elevations of SGPT (ALT) or SGOT (AST) greater than 2 1/2 times normal at screening.
11. Females of child bearing potential who are pregnant (by urine HCG), nursing, or who are not using a reliable form of birth control.
12. Has current charges pending for a violent crime (not including DUI related offenses).
13. Does not have a stable living situation.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160
Dates: Start 2005-05; Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
"Natural" alcohol consumption period -- Total number of drinks consumed during the 5 day observation period
Pharmacological effects of alcohol consumption -- Average BAES stimulation score
Limited access alcohol consumption paradigm -- Total number of drinks consumed
Cue induced brain imaging -- Alcohol beverage cue minus neutral beverage cue activity in nucleus accumbens and insula

SECONDARY OUTCOMES:
Change in craving as measured by the OCDS from pre-study to end of 5 day period
Change in craving from pre to post-alcohol ingestion
Change in craving during limited-access alcohol consumption
Change in craving during cue-induced brain activity
Side effects of medications

CONTACTS AND LOCATIONS:
Overall Officials: Raymond F Anton, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Center for Drug and Alcohol Programs, Medical University of South Carolina, Charleston, South Carolina, United States